CLINICAL TRIAL: NCT06176170
Title: A Prospective Multicentre Pivotal Clinical Study to Demonstrate the Efficacy and Safety of the VividWhite Glaucoma Implant (VW-51) for the Treatment of Glaucoma.
Brief Title: VividWhite Glaucoma Implant (VW-51) Pivotal Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VividWhite Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DF-550
Record Dates: First submitted 2023-12-10; First posted 2023-12-19 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VividWhite Glaucoma Implant (VW-51) (Experimental): Surgical implantation of VW-51.
  Interventions: Device: VividWhite Glaucoma Implant (VW-51)

INTERVENTIONS:
Device: VividWhite Glaucoma Implant (VW-51) — Subconjunctival surgical implantation of the VW-51 implant in the study eye.

SUMMARY:
The VividWhite Glaucoma Implant (VW-51) is a novel surgical implant designed to treat glaucoma. This study is a 12-month, 65-participant non-comparative multicentre study to assess the safety and effectiveness of the VW-51 implant.

DETAILED DESCRIPTION:
A prospective multicentre non-comparative pivotal clinical study where all participants undergo treatment with a novel surgical implant (VW-51) and receive 12 months of clinical follow-up. The study aim is to assess the effectiveness, safety and participant experience of the VW-51 implant for the treatment of glaucoma. The study population will involve 65 adult participants with medically or surgically refractory glaucoma. The VW-51 implant is a leaf-shaped microfluidic device manufactured from flexible silicone, designed to be surgically implanted in the subconjunctival space, drain aqueous humor from the eye and reduce intraocular pressure to treat glaucoma.

ELIGIBILITY:
Key Inclusion Criteria: Glaucoma in the study eye, meeting the following requirements:

1. Glaucoma is diagnosed by the investigator based upon untreated intraocular pressure, disc appearance and visual field abnormalities, and where the disease type is one of: Primary open angle glaucoma (POAG); Chronic angle closure glaucoma (CACG) where the eye is pseudophakic and a laser iridotomy has previously been performed; Pigmentary open angle glaucoma; Exfoliation open angle glaucoma; Rubeotic glaucoma that is treated and regressed/quiescent; Steroid-induced glaucoma; or Juvenile open angle glaucoma (JOAG).
2. There has been failure of previous treatment for glaucoma (it is 'refractory'), meeting ONE of the following requirements:

i. Failure of medical treatment: inadequate IOP control on maximum tolerated medical therapy.

ii. Failure of previous glaucoma surgery (not more than one operation) with trabeculectomy, Xen/PreserFlo, non-penetrating glaucoma surgery, a previously removed suprachoroidal drainage device, trabecular bypass (using iStents or Hydrus), or cilioablation.

c. The mean diurnal IOP at Screening/Baseline is ≥ 20 mmHg, and ≤ 40 mmHg.

d. The conjunctiva in the target quadrant is healthy, mobile and suitable for glaucoma surgery.

Key Exclusion Criteria: in the study eye:

1. Advanced glaucomatous optic neuropathy that threatens fixation, in the opinion of the investigator.
2. The glaucoma type is any of the following: Acute Angle Closure Glaucoma (AACG); Chronic Angle Closure Glaucoma where the eye is phakic; Congenital glaucoma; or Secondary glaucoma of any type not specified in the inclusion criteria, including inflammatory glaucoma, active neovascular/rubeotic glaucoma, traumatic glaucoma, Iridocorneal Endothelial (ICE) Syndrome, and silicone oil induced glaucoma.
3. Previous glaucoma surgery with: a tube-and-plate glaucoma drainage device (GDD, e.g. Molteno, Baerveldt, Ahmed, Schocket); an in-situ suprachoroidal implant; or multiple previous operations for glaucoma.
4. Cataract surgery or any other ocular surgery is indicated at the time of study intervention or is anticipated to be required during the study duration.
5. Central corneal endothelial cell density less than specified age-related thresholds at screening.
6. Intraocular silicone oil.
7. Significant corneal, retinal, inflammatory or infective ophthalmic pathology (full details specified in the protocol).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Complete success by efficacy and safety criteria | Study completion (12 months)
  Efficacy Criteria:
  1. Intraocular pressure (IOP) is less than or equal to 21 mmHg.
  2. IOP is reduced by greater than or equal to 20% compared to baseline (mean diurnal).
  3. Treatment with the same number or fewer classes of topical glaucoma medication than at baseline.
  4. No requirement for: further glaucoma surgery indicated for efficacy (at any time during the study); or systemic/oral ocular hypotensive medication to achieve target IOP in the study eye (at any time during the study).
     Safety Criteria:
  5. IOP is greater than or equal to 6 mmHg.
  6. No adverse events of special significance in the study eye (as specified by the protocol; for example further glaucoma surgery indicated for safety).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Coote, Principal Investigator — Melbourne Eye Specialists
Locations (6):
- Australia (6):
  - Sydney Eye Hospital, Sydney, New South Wales
  - Flinders Medical Centre, Bedford Park, South Australia
  - Cataract & Eye Surgery Centre, Doncaster East, Victoria
  - Cerulea Clinical Trials, Centre for Eye Research Australia, East Melbourne, Victoria
  - Melbourne Eye Specialists, Fitzroy, Victoria
  - Eye Surgery Associates, Vermont South, Victoria

IPD SHARING:
Plan to Share IPD: No